(De- Escalation and Stopping Treatment of Imatinib, Nilotinib or sprYcel in chronic myeloid leukaemia) (DESTINY)

NCT01804985

ISRCTN Number: 74084226

EudraCT number: 2012-004025-24

Final Statistical Analysis Report Plan

Version 1

17<sup>th</sup> July 2019







A trial of de-escalation and stopping treatment in chronic myeloid leukaemia patients with excellent responses to tyrosine kinase inhibitor therapy

(De- Escalation and Stopping Treatment of Imatinib, Nilotinib or sprYcel in chronic myeloid leukaemia)
(DESTINY)

ISRCTN Number: 74084226

EudraCT number: 2012-004025-24

# Final Statistical Analysis Report Plan

Prepared by: Silvia Cicconi - Trial Statistician

# Contents

| 1. | INTRODUCTION | 4 |
|----|-----------------------------------------------------|--------------|
| 2. | TRIAL DESIGN | 5 |
| | 2.1. Configuration | 5 |
| | 2.2. Interventions | 5 |
| | 2.3. Objectives | 5 |
| | 2.4. Eligibility Criteria | 5 |
| | 2.5. Sample size | 6 |
| | 2.6. Randomisation procedure | 6 |
| | 2.7. Blinding | 6 |
| | 2.8. Endpoints | 7 |
| | 2.9. Interim Monitoring and Analyses | 7 |
| 3. | TRIAL HISTORY | 9 |
| | 3.1. Quality control and data validation procedures | 9 |
| | 3.2. Protocol Amendments | 9 |
| | 3.3. Trial Milestones | 9 |
| 4. | PROPOSED METHODOLOGY | 0 |
| | 4.1. Patient Groups for Analysis | . 10 |
| | 4.2. Handling of dropouts | . 10 |
| | 4.3. Identification and handling of Outliers | . 10 |
| | 4.4. Study centre effects | . 11 |
| | 4.5. Adjustment for covariates | . 11 |
| | 4.6. Multiplicity adjustments | . 11 |
| | 4.7. Missing data | . 11 |
| | 4.8. Sensitivity analyses | . 11 |
| | 4.9. Pre-specified subgroup analyses | . 11 |
| | 4.10. Derived variables & Definitions | . 12<br>. 12 |
| | 4.11. Null hypothesis, levels of significance | . 14 |

| 5.1. Recruitment and disposition | ESULTS | 16 |
|---|---|---|
| 5.3. Description of baseline subject characteristics 20 5.4. Exposure to treatment and compliance 22 5.5. Analysis of Primary Outcome 22 5.6. Analyses of secondary outcomes 22 Relapse on cessation 22 Regained MMR 22 Molecular relapse-free survival 22 Progression-free Survival 22 Overall Survival 22 Event-free survival 22 Time to MMR recovery 22 MR <sup>4.5</sup> prior study entry 22 Quality of Life and TKI related symptoms 22 | .1. Recruitment and disposition | 16 |
| 5.4. Exposure to treatment and compliance | .2. Assessment of data quality | 18 |
| 5.5. Analysis of Primary Outcome | .3. Description of baseline subject characteristics | 20 |
| 5.6. Analyses of secondary outcomes 22 Relapse on cessation 22 Regained MMR 22 Molecular relapse-free survival 22 Progression-free Survival 22 Overall Survival 22 Event-free survival 22 Time to MMR recovery 22 MR <sup>4.5</sup> prior study entry 29 Quality of Life and TKI related symptoms 29 | .4. Exposure to treatment and compliance | 21 |
| Relapse on cessation | .5. Analysis of Primary Outcome | 21 |
| Progression-free Survival 25 Overall Survival 26 Event-free survival 27 Time to MMR recovery 25 MR <sup>4.5</sup> prior study entry 29 Quality of Life and TKI related symptoms 29 | Relapse on cessation | 22<br>23 |
| Time to MMR recovery | Progression-free Survival Overall Survival | 25<br>26 |
| | Time to MMR recoveryMR <sup>4.5</sup> prior study entry | 28<br>29 |

#### 1. INTRODUCTION

This document details the rules proposed and the presentation that will be followed, as closely as possible, when analysing and reporting the main results from the trial of deescalation and stopping treatment in chronic myeloid leukaemia funded by the Leukaemia and Lymphoma Research Clinical Trials Committee.

The purpose of the plan is to:

- a. Ensure that the analysis is appropriate for the aims of the trial, reflects good statistical practice in general, and minimises bias by preventing inappropriate post hoc analyses;
- b. Explain in detail how the data will be handled and analysed to enable others to perform the actual analysis in the event of sickness or other absence;
- c. Protect the project by helping it keep to timelines and within scope.

Additional exploratory or auxiliary analyses of data not specified in the protocol are permitted but fall outside the scope of this analysis plan (although such analyses would be expected to follow Good Statistical Practice).

The analysis strategy will be made available if required by journal editors or referees when the main papers are submitted for publication. Additional analyses suggested by reviewers or editors will, if considered appropriate, be performed in accordance with the Analysis Plan, but if reported the source of such a post-hoc analysis will be declared.

Amendments to the statistical analysis plan will be described and justified in the final report of the trial.

#### 2. TRIAL DESIGN

#### 2.1. Configuration

A multi-centre, single arm, Phase II, prevalence study.

### 2.2. Interventions

De-escalation to half the standard TKI dose for up to 13 months, followed by 2 years treatment cessation. If on imatinib, the dose should be decreased to 200mg daily; if on nilotinib to 200mg twice daily and if on dasatinib to 50 mg daily.

## 2.3. Objectives

To determine the safety and efficacy of initially de-escalating and then stopping TKI treatment, in CML patients with either undetectable disease or with stable MMR.

## 2.4. Eligibility Criteria

#### **Inclusion Criteria**

- 1. CML in first chronic phase.
- 2. Demonstration of BCR-ABL1 positivity at or shortly after original diagnosis\*.
- 3. Written Informed Consent
- 4. Must have received TKI treatment for at least 3 years.
- 5. At least 3 molecular results over the preceding 12 months that fit either of the following groups (results from any UK lab are acceptable):
  - (MR<sup>4</sup> group) all the available BCR-ABL1 molecular results over the preceding 12 months are in MR<sup>4</sup> (MR<sup>4</sup> is defined as a BCR-ABL1/ABL1 ratio of zero, (reported to international standard (IS) where possible); with at least 10,000 ABL1 control transcripts).
  - (MMR group) some or all BCR-ABL1 molecular results are in MMR (BCR-ABL1/ABL1 ratio of 0.1% or less, (reported to International Standard (IS) where possible), but not zero, with at least 10,000 ABL1 control transcripts). If the results over the preceding 12 months are a mix of MMR and undetectable BCR-ABL1, then the patient is eligible for the MMR but not the MR<sup>4</sup> group.

#### **Exclusion Criteria**

- 1. Age under 18
- 2. Life expectancy is predicted to be less than 37 months because of intercurrent illness
- 3. Presence of serious concomitant illness (e.g. heart, renal, respiratory or active malignant disease) that might preclude completion of the trial
- 4. CML in accelerated phase or blast crisis at any time
- 5. Any molecular result during the preceding 12 months that is not in either MMR or MR<sup>4</sup>.

<sup>\*</sup> Patients who are Philadelphia chromosome (Ph) negative (or whose Ph status is not known) are eligible. Patients who do not have a standard BCR-ABL1 fusion transcript (i.e. other than e13a2 or e14a2, also known as b2a2 and b3a2) may be eligible, but before screening the patient, contact should be made with Prof Foroni at Hammersmith Hospital (see contacts in the Protocol) since specialised quantitative molecular assessment will be required.

- 6. Patients who switched previous licensed TKI treatment (imatinib, nilotinib or dasatinib) twice or more because of intolerance.
- 7. Treatment with higher than standard TKI doses ('standard' is defined as imatinib 400mg daily, nilotinib 400mg twice daily or dasatinib 100mg daily). However, an exception is made for patients who at original diagnosis commenced on either 800mg of imatinib on the SPIRIT1 study, or 140mg (or 70mg b.d.) of dasatinib in the Bristol-Myers Squibb 034 study. In each case these latter patients ARE eligible provided they fulfil other molecular criteria, since they do not demonstrate resistant disease.
- 8. Patients who switched previous licensed TKI treatment (imatinib, nilotinib or dasatinib) because of resistance. Patients treated with lower (but at least 50%) than standard TKI doses (as defined in the previous criterion) for tolerance reasons may be included, but will de-escalate to the same doses as for standard dose patients and will be analysed separately, as they could be seen as undertreated.
- 9. Previous treatment with ponatinib or bosutinib. Patients who received interferon prior to commencing TKI (even if resistant to their interferon) are eligible, provided their response to TKI fits the entry criteria and the use of interferon ceased at least 12 months prior to study entry.
- 10. Pregnant or lactating women
- 11. Women of childbearing potential, including women whose last menstrual period was less than one year prior to screening, unable or unwilling to use adequate contraception from trial start to one year after the last dose of protocol therapy. Adequate contraception is defined as hormonal birth control, intrauterine device, double barrier method or total abstinence.

#### 2.5. Sample size

Seventy cases will give a 90% confidence interval of maximum width 0.2, for a wide range (0.3 to 0.7) of values of the proportion, p, of relapsing patients. The width will be smaller the closer the estimate is to 0 (or 1). Assuming a dropout rate of 17% and an anticipated equal group allocation, 168 patients are needed.

The accrual of patients within each group largely depends on factors that cannot be controlled or specified a-priori. Hence, to avoid early closing of recruitment in one group which could potentially have a negative effect in overall recruitment and would require substantial extension in the recruitment period we are willing to allow for unequal group allocation and some variation in the maximum confidence interval width. Assuming that we recruit 168 patients in total, under the worst case scenario (p=0.5, group allocation 1:3) the 90% confidence intervals for the two groups ("larger" and "smaller") will have a maximum width of 0.16 and 0.28 respectively.

#### 2.6. Randomisation procedure

None – this is a single arm trial.

## 2.7. Blinding

None - open label

#### 2.8. Endpoints

#### **Primary outcome**

The proportion of patients who can first de-escalate their treatment (to half the standard dose of their TKI) for 12 months, and then stop treatment completely for a further 2 years, without losing MMR. This will be calculated separately for each of the two groups (MR<sup>4</sup> and MMR).

#### **Secondary outcomes**

- Proportion of patients who can successfully de-escalate their treatment (to half the standard dose of their TKI), but who then lose MMR on complete TKI cessation.
- Proportion of patients who lose their MMR on de-escalation/stopping and regain MMR on resumption of their TKI.
- Molecular relapse-free survival (RFS); RFS is defined as the time from the first day of deescalation to the date of confirmed loss of MMR (two consecutive BCR-ABL >0.1% IS).
- Progression-free survival (PFS); PFS is defined as the time from the first day of deescalation to the date of progression to accelerated phase/ blast crisis or death from any cause (earliest occurrence).
- Overall survival (OS); OS is defined as the time from the first day of de-escalation to the date of death from any cause.
- Event-free survival (EFS); EFS is defined as the time from the first day of de-escalation to the date of confirmed loss of MMR, progression to AP/BC or death from any cause.
- Time to MMR recovery (TTR); TTR is defined as the time from the date of confirmed loss of MMR to the date of MMR recovery.
- Proportion of registered MMR and MR<sup>4</sup> patients in confirmed MR<sup>4.5</sup> (BCR-ABL ≤ 0.0032% IS with at least 31,623 ABL1 control transcripts) prior to being enrolled in the study (screening phase).
- · Quality of Life
- Health Economic Assessment
- Lab studies to define subsets of patients who are more likely to relapse on de-escalation / cessation.

The last two secondary outcomes are not part of this statistical analysis plan.

#### 2.9. Interim Monitoring and Analyses

The proportion of relapsing patients will be assessed at 3 planned interim analyses: when 60 patients relapse or complete 12 months de-escalation, when 60 relapse or complete 12 months of cessation, and when 60 relapse or complete 24 months cessation. There are no formal stopping rules but the Independent Data Monitoring and Safety Committee (ISDMC) will review the interim analyses and give advice on whether the accumulated data from the trial, together with results from other relevant trials, justifies continuing recruitment of further patients or further follow-up.

A decision to discontinue recruitment will be made only if the result is likely to convince a broad range of clinicians including participants in the trial and the general clinical community. The entire trial (or the MMR or MR<sup>4</sup> elements alone) may be stopped if de-escalation or

stopping are producing an unacceptable rate of molecular relapse. For this purpose, the MMR and  $MR^4$  groups will be treated separately, since the former may well have a higher relapse rate. Unacceptable relapse for this purpose is at the discretion of the Data Monitoring Committee, bearing in mind that the relapse rate in the STIM trial was 61% overall and 59% (48% - 71%) after 12 months of cessation.

Regardless of the reason(s) for termination, all data available for the patient at the time of discontinuation of follow-up must be recorded in the CRF. All reasons for discontinuation of treatment must be documented. In terminating the trial, the sponsor and the Investigators will ensure that adequate consideration is given to the protection of the patient's interest.

All interim analysis results of the primary and secondary outcome measures will be confidential to the ISDMC members and will not be for review by the trial management group (except the trial statistician preparing the ISDMC report), Trial Steering Committee, investigators or collaborators.

#### 3. TRIAL HISTORY

## 3.1. Quality control and data validation procedures

#### Randomisation checks

Not applicable – there is no randomisation in this trial.

## Derivation of primary outcome

The code for derivation of the primary outcome will be validated by an independent statistician on a risk approach basis. The same will apply to secondary outcomes code.

#### **Automated checks**

The MACRO database includes validation features which to alert the user to certain inconsistent or missing data on data entry and automatically raise a query which is emailed to the research site. Automated email reminders are also generated by the database if follow up data from a scheduled patient visit is overdue.

#### Other checks

Eligibility criteria, informed consent and registration dates/numbers are checked by the trial team at the time of registration.

#### 3.2. Protocol Amendments

This will include a short summary of all protocol amendments.

#### 3.3. Trial Milestones

| First patient was recruited on: |
|------------------------------------------------|
| Latest patient was recruited on: |
| Cut-off date (data freeze) for this report: |
| Date of final data extraction for this report: |
| Total number screened to data freeze: |
| Total number recruited to data freeze: |
| Target number of patients: |
| Proportion of target number recruited: |

#### 4. PROPOSED METHODOLOGY

The trigger for the final analysis will be the date when the last relapse-free patient completes 37 months of follow-up or the date when the last relapsed patient regains MMR (latest occurrence) unless the TSC decides to terminate the trial prematurely.

As this is a prevalence study, analyses of the two cohorts (MMR and MR<sup>4</sup>) will be carried out separately, using the same methods for each. For any statistical analysis MR<sup>4</sup> patients will be re-classified to either MMR or MR<sup>4</sup> group based on the following criterion:

• MR<sup>4</sup>: At least complete molecular remission MR<sup>4</sup> (either (i) detectable disease ≤0.01% BCR-ABL IS or (ii) undetectable disease in cDNA with ≥ 10,000 ABL or ≥ 24,000 GUS transcripts) for at least one year; at least three PCR-results with MR<sup>4</sup> within the last year (+- 2 months) before study entry and no PCR-results > 0.01% during the same period.

#### 4.1. Patient Groups for Analysis

<u>Full Analysis set</u>: In order to follow the Intention to Treat (ITT) principle this consists of all registered patients excepting for:

- a) Patients withdrawing consent between registration and starting therapy
- **b)** Patients withdrawn from the study after registration because of irregularities with the consent process and
- **c)** Patients whose information determining ineligibility existed before registration but was not read until after registration.

<u>Per protocol set</u>: This consists of those patients in the Full Analysis set without any major protocol deviations, following review by the Trial Management Group.

**<u>Safety set</u>**: All patients who received any trial treatment.

#### 4.2. Handling of dropouts

Dropouts, that is unevaluable patients, will be censored at last visit date in survival analyses or treated as non-responders for the purpose of clinical response.

#### 4.3. Identification and handling of Outliers

For continuous variables potential outliers will be defined as follows (Tukey, 1977)<sup>1</sup> after testing for symmetry and if non-symmetric, transforming to approximate symmetry using a "ladder of powers" approach using the Stata command *ladder*:

"Mild" outliers: UQ+1.5×IQR to UQ+3×IQR or LQ-1.5×IQ to LQ-3×IQR

"Severe" outliers: values more extreme than the above

(Note: UQ=Upper Quartile, LQ=Lower Quartile, IQR=Inter Quartile Range)

If after transformation no outliers are apparent then no action will be taken even if values appear as outliers on the original scale, apart from use of the transformation if normality is

<sup>&</sup>lt;sup>1</sup> Tukey, J.W. (1977), Exploratory Data Analysis, Reading, MA: Addison-Wesley

required for a particular statistical procedure, or to remove the leverage effect of the outlying values.

Otherwise outliers in quantitative data will be queried but no action taken if the result is not amended.

#### 4.4. Study centre effects

There will be limited capacity to investigate these formally and such centre effects are to be expected by chance.

## 4.5. Adjustment for covariates

No appropriate adjustment for covariates has been identified.

## 4.6. Multiplicity adjustments

No adjustment will be made.

## 4.7. Missing data

This problem is not expected to arise for the primary outcome analysis; the primary outcome is relapse rate which is easily ascertained. If >20% of patients have missing/unacceptable values on any of the variables of interest (e.g., secondary outcomes), then multiple imputation should be attempted, performing at least 10 separate sets of multiple imputations using chained equations using separate imputations for MMR and MR<sup>4</sup> groups.

#### 4.8. Sensitivity analyses

These will consist of:

• Per-protocol analysis for primary endpoint

## 4.9. Pre-specified subgroup analyses

The final analysis of primary and secondary outcomes will be analysed in the following subgroups:

- MMR
- MR<sup>4</sup>

The primary outcome and time to molecular relapse will also be analysed according to MR<sup>4.5</sup> status prior entering the study within each subgroup:

- MMR MR<sup>4.5</sup>
- MMR not MR<sup>4.5</sup>
- MR<sup>4</sup> MR<sup>4.5</sup>
- MR<sup>4</sup> not MR<sup>4.5</sup>

#### 4.10. Derived variables & Definitions

#### **Definitions**

**Cut-off date**: this is the date after which all events, readings etc. are ignored, in order to provide a defined reference point for calculating survival time, etc. For the final analysis the cut-off date will be the date of completion of minimum follow-up on last patient.

**Exit date**: this is the date assigned to the event of interest (progression, death, etc.) provided this is earlier than the cut-off date. If date of event is known to be later than the cut-off date then the exit date = cut-off date. If date of event is not recorded then the exit date will be the most recent visit date.

*Visit date*: this is the date of patient attendance for assessment, treatment etc.

**Exit status**: this is coded as "1" if the event of interest has occurred, "0" otherwise (censoring indicator).

## **Primary Outcome**

 Proportion of patients who can first de-escalate their treatment (to half the standard dose of their TKI) for 12 months, and then stop treatment completely for a further 2 years, without losing MMR.

Event of interest = Molecular Relapse by the end of month 37 - defined as loss of MMR on 2 consecutive occasions (BCT-ABL > 0.1% IS)

Relapse date = the date that the confirmation sample was collected

## **Secondary outcomes**

 Proportion of patients who can successfully de-escalate their treatment (to half the standard dose of their TKI), but who then lose MMR on complete TKI cessation.

Event of interest = Molecular Relapse after 12 months of de-escalation
Relapse date = the date that the confirmation sample was collected
Exit date = Relapse date if Relapse date < cut-off date, last visit date otherwise

 Proportion of patients who lose their MMR on de-escalation/stopping and regain MMR on resumption of their TKI.

Event of interest = Regaining MMR after relapse
Regaining MMR date = the date that the confirmation sample was collected
Exit date = Regain MMR date if Regain MMR date < cut-off date, last visit date otherwise

Molecular relapse-free survival (RFS).

RFS is defined as the time from the first day of de-escalation to the date of confirmed loss of MMR (two consecutive BCR-ABL > 0.1% IS).

Date of event = Date of confirmed loss of MMR

Exit date = Date of confirmed loss of MMR if date < cut-off date, last visit date otherwise  $Relapse-free\ Survival\ (months) = \{exit\ date - date\ of\ first\ day\ of\ de-escalation\}/30.4$ 

Exit status = 1 if molecular relapse occurred before cut-off date, 0 otherwise

## • Progression-free survival

PFS is defined as the time from the first day of de-escalation to the date of progression to accelerated phase/blast crisis or death from any cause (first occurrence).

Event of interest = progression to accelerated phase/blast crisis

Progression date = min( date of death, Progression date)

Exit date = Progression date if Progression date < cut-off date, last visit date otherwise Progression-free Survival (months) = (exit date – date of first day of de-escalation)/30.4 Exit status = 1 if disease progression or dead from any cause before cut-off date, 0 otherwise.

#### • Overall survival

OS is defined as the time from the first day of de-escalation to the date of death from any cause.

Event of interest = death from any cause

Date of event = Date of death

Exit date = Date of death if date < cut-off date, last visit date otherwise

Overall Survival (months) = {exit date - date of first day of de-escalation}/30.4

Exit status = 1 if dead before cut-off date, 0 otherwise

# • Event-free survival (EFS)

EFS is defined as the time from the first day of de-escalation to the date of confirmed loss of MMR, progression to AP/BC or death from any cause.

Date of event = Date of EFS event

Exit date = Date of EFS event if date < cut-off date, last visit date otherwise Event-free Survival (months) = {exit date – date of first day of de-escalation}/30.4 Exit status = 1 if event occurred before cut-off date, 0 otherwise

## • Time to MMR recovery (TTR)

TTR is defined as the time from the date of confirmed loss of MMR to the date of MMR recovery.

Date of event = Date of MMR recovery

Exit date = Date of MMR recovery if date < cut-off date, last visit date otherwise

TTR (months) = {exit date - date of confirmed loss of MMR}/30.4

Exit status = 1 if MMR recovery occurred before cut-off date, 0 otherwise

Proportion of registered MMR and MR<sup>4</sup> patients in confirmed MR<sup>4.5</sup> (BCR-ABL ≤ 0.0032% IS with at least 31,623 ABL1 control transcripts) prior to being enrolled in the study (screening phase).

 $MR^{4.5}$  is defined as MMR or  $MA^4$  patients with BCR-ABL  $\leq 0.0032\%$  IS and at least 31,623 ABL1 control transcripts prior to entering the study.

# Quality of life

Quality of life will be assessed using the EQ-5D, EQ-VAS and FACT-BRM questionnaires. Additional information collected regarding TKI related symptoms will also be assessed.

# 4.11. Null hypothesis, levels of significance

Since this is a prevalence study the aim is to provide estimates of the efficacy parameters with a certain level of confidence. The primary efficacy parameter of relapse rate will be estimated on an Intention-to-Treat basis and reported together with a 90% confidence interval. All secondary parameter estimates will also be reported with 90% confidence intervals.

# 4.12. Specification and estimation of efficacy parameters

Table 1: Summary of outcome variables and corresponding efficacy parameters.

| Outcome variable | Efficacy parameter | Comment | Method |
|---|---|---|---|
| Relapse rate | Proportion of patients with<br>molecular relapse at any<br>time point during the 37<br>months | Estimated separately for<br>each cohort (MMR, MR <sup>4</sup> ) and<br>for the MR <sup>4.5</sup> subgroups<br>(MMR-MR <sup>4.5</sup> , MMR-<br>notMR <sup>4.5</sup> , MR <sup>4</sup> -MR <sup>4.5</sup> , MR <sup>4</sup> -<br>notMR <sup>4.5</sup> ) | Binomial proportion with normal approximation confidence interval |
| Relapse rate after<br>successful de-<br>escalation | Proportion of patients with molecular relapse after successful de-escalation | Estimated separately for each cohort (MMR, MR <sup>4</sup> ) | Binomial proportion with normal approximation confidence interval |
| Regain MMR rate | Proportion of patients who regain MMR after molecular relapse at any time point | Estimated separately for each cohort (MMR, MR <sup>4</sup> ) | Binomial proportion with normal approximation confidence interval |
| Molecular Relapse-<br>free survival (RFS) | Median RFS time | Supported by • 12-36 months RFS Estimated separately for each cohort (MMR, MR <sup>4</sup> ) and for the MR <sup>4.5</sup> subgroups (MMR-MR <sup>4.5</sup> , MMR-notMR <sup>4.5</sup> , MR <sup>4</sup> -MR <sup>4.5</sup> , MR <sup>4</sup> -notMR <sup>4.5</sup> ) | Kaplan-Meier<br>estimator with<br>pointwise bounds |
| Progression-free<br>Survival (PFS) | Median PFS time | Supported by • 12-36 month PFS Estimated separately for each cohort (MMR, MR <sup>4</sup> ) | Kaplan-Meier<br>estimator with<br>pointwise bounds |
| Overall survival<br>(OS) | Median OS time | Supported by • 12-36 month OS Estimated separately for each cohort (MMR, MR <sup>4</sup> ) | Kaplan-Meier<br>estimator with<br>pointwise bounds |

| Event-free survival | Median EFS time | Supported by | Kaplan-Meier |
|---|---|---|---|
| (EFS) | | • 12-36 month EFS | estimator with |
| | | | pointwise bounds |
| | | Estimated separately for | |
| | | each cohort (MMR, MR <sup>4</sup> ) | |
| Time to MMR | Median TTR time | Supported by | Cumulative |
| recovery (TTR) | | • 12-36 month TTR | incidence estimate |
| | | | adjusting for the |
| | | Estimated separately for | competing risks of |
| 4.5 | | each cohort (MMR, MR <sup>4</sup> ) | progression/death |
| MR <sup>4.5</sup> rate | Proportion of MMR and | Estimated separately for | Binomial proportion |
| | MR <sup>4</sup> patients in confirmed | each cohort (MMR, MR <sup>4</sup> ) | with normal |
| | MR <sup>4.5</sup> prior to entering the | | approximation |
| | study | | confidence interval |
| Quality of Life | Mean scores at baseline | Estimated separately for | Graphs showing |
| | and each time point | each cohort (MMR, MR <sup>4</sup> ) | measurements |
| | questionnaires were | | overtime. Further |
| | completed | | QoL assessments |
| | | | will be performed |
| | | | using joint |
| | | | longitudinal and |
| | | | survival analysis to |
| | | | assess the |
| | | | difference between |
| | | | relapsing and not |
| | | | relapsing patients |

# **5. RESULTS**

# 5.1. Recruitment and disposition

**Table 2: Recruitment by centre** 

| Site Name | Date of green light* | Date of first recruitment | Date of last recruitment | MMR | MR <sup>4</sup> | Total |
|---|---|---|---|---|---|---|
| | | | Total | | | |

Figure 1: Recruitment graph (example)



Figure 2: Patient disposition



# 5.2. Assessment of data quality

**Table 3: Protocol treatment & Trial dropouts** 

| | MMR | MR⁴ | Overall |
|---|---|---|---|
| Characteristic | N = | N = | N = |
| Total discontinued protocol treatment [n, (%)] | | | |
| Serious Adverse Event/ Toxicity | | | |
| Death | | | |
| Patient / Clinical decision (not SAE, not trial related) | | | |
| Serious violation of study protocol | | | |
| Withdrawal of consent | | | |
| Disease progression/ Molecular Relapse | | | |
| Intercurrent illness | | | |
| Other | | | |
| Reason missing | | | |
| Days from recruitment to discontinuation of | | | |
| protocol <u>treatment</u> | | | |
| Median | | | |
| IQR | | | |
| Range | | | |
| Total discontinued <u>trial</u> [n, (%)] | | | _ |
| Consent withdrawn | | | |
| Lost to follow up | | | |
| Death | | | |
| Other | | | |
| Days from recruitment to discontinuation of trial | | | |
| Median | | | |
| IQR | | | |
| Range | | | |

**Protocol deviations**: Protocol Deviations are accidental or unintentional change to or noncompliance with the trial protocol.

**Table 4a: Summary of Deviations** 

| Туре | Description of Deviation | Category | Total No. |
|---|---|---|---|
| | Entered but subsequently found not to satisfy the entry criteria | 1 | |
| | Developed withdrawal criteria but not withdrawn | 2 | |
| Major | Received an excluded concomitant treatment | 3 | |
| | Received the wrong treatment or incorrect dose | 4 | |
| | Deviation from patient management/assessment | 5 | |
| | Other | 6 | |

| Minor | Protocol Deviations not expected to have an | 7 |
|----------|---------------------------------------------|---|
| IVIIIIOI | impact on defined endpoints of the trial | , |

Review for Major Deviations will be performed by the Trial Management Group on a regular basis (hence before any per-protocol analysis).

Table 4b: Details of Major Deviations by site

| Site Name | Date | Category | Details |
|-----------|------|----------|---------|

**Table 5: Available Data Description** 

| Patients missing values on: | MMR | MR <sup>4</sup> |
|------------------------------|-----|-----------------|
| Primary outcome | | |
| Relapse Rate | | |
| Secondary outcomes | | |
| Relapse rate after 12 months | | |
| Regain MMR rate | | |
| Relapse-free Survival | | |
| Progression-free Survival | | |
| Overall Survival | | |
| Event-free Survival | | |
| Time to MMR recovery | | |

# **5.3.** Description of baseline subject characteristics

Categorical variables are summarised as N (%); continuous variables by mean (SD) and lower and upper quartiles.

**Table 6: Baseline characteristics** 

| Table 6: Baseline Characteristics | MMR | MR <sup>4</sup> | Overall |
|---|---|---|---|
| | N = | N = | N = |
| Demographic Characteristics | | | 1 |
| Age | | | |
| median (IQR) | | | |
| Gender [n (%)] | | | |
| Male | | | |
| Female | | | |
| Physical findings | | | 1 |
| Weight | | | |
| median (IQR) | | | |
| ECOG performance status [n, (%)] | | | |
| Fully Active | | | |
| Work Able | | | |
| Not Work Able | | | |
| Limited Self Care | | | |
| Completely Disabled | | | |
| Clinical characteristics | | | 1 |
| BCR-ABL % (Hammersmith results) | | | |
| median (IQR, range) | | | |
| Medical History | | | |
| Medical history or baseline symptoms [n (%)] | | | |
| None | | | |
| Current<br>Previous | | | |
| Medication | | | |
| Current CML Medication [n (%)] | | | |
| Imatinib | | | |
| Nilotinib | | | |
| Dasatinib | | | |
| Haematology results | | | 1 |
| Haemoglobin g/L | | | |
| median (IQR) | | | |
| WBC ×10 <sup>9</sup> | | | |
| median (IQR) | | | |
| TKI related symptoms | | l | I |
| Symptom [n, (%)] | | | |
| Rash | | | |
| Diarrhoea | | | |
| Nausea<br>Scala irritation | | | |
| Scalp irritation Periobital oedema | | | |
| Hair thinning | | | |
| Lethargy<br>Other | | | |
| Other | | | l |

| Grade CTCAE [n, (%)] | |
|----------------------|----|
| | 3+ |
| | <3 |

# 5.4. Exposure to treatment and compliance

Table 7: Details of treatment doses administered

| Group | No. of patients<br>administered at<br>least one day of<br>protocol<br>treatment | No. of patients<br>with at least<br>one dose<br>missed | No. of patients with at least one dose increase | No. of patients with premature TKI cessation |
|---|---|---|---|---|
| MMR | | | | |
| MR <sup>4</sup> | | | | |

# 5.5. Analysis of Primary Outcome

**Table 8: Relapse rate at 37 months** 

| Group | Total no. of patients | No. of evaluable patients * | Completeness<br>of follow up<br>(C) <sup>2</sup> | No. of relapsed patients | % of evaluable patients who completed 37 months without relapse | 90%<br>Confidence<br>Interval |
|---|---|---|---|---|---|---|
| MMR | | | | | | |
| MR <sup>4</sup> | | | | | | |

<sup>\*</sup>Subtracting losses to follow-up & complete withdrawals (prior to experiencing any event) from the total.

 $^2$  Clark TG, Altman DG, De Stavola BL (2002) "Quantification of the completeness of follow-up" Lancet 359: 1309-1310

Table 9: Results of Sensitivity analyses for relapse rate at 37 months

| Sensitivity<br>Analysis -<br>allowance for | Group | No. of patients | No. of<br>evaluable<br>patients | No. of relapsed patients | % of evaluable patients<br>who completed 37<br>months without<br>relapse | 90 %<br>Confidence<br>Interval |
|---|---|---|---|---|---|---|
| Per-protocol | MMR | | | | | |
| analysis | MR <sup>4</sup> | | | | | |

# Table 10: Results of subgroup analysis based on MR<sup>4.5</sup> status for relapse rate at 37 months

| Group | No. of patients | No. of<br>evaluable<br>patients | No. of relapsed patients | % of evaluable patients who completed 37 months without relapse | 90 %<br>Confidence<br>Interval |
|---|---|---|---|---|---|
| MMR – MR <sup>4.5</sup> | | | | | |
| MMR – not MR <sup>4.5</sup> | | | | | |
| MR <sup>4</sup> – MR <sup>4.5</sup> | | | | | |
| MR <sup>4</sup> – not MR <sup>4.5</sup> | | | | | |

# **5.6.** Analyses of secondary outcomes

# Relapse on cessation

Table 11: Results for patients who relapse on cessation

| Group | No. of patients | No. of patients who completed de-escalation without relapsing | No. of relapsed patients after de-escalation | % of patients<br>who relapse<br>on cessation | 90%<br>Confidence<br>Interval |
|---|---|---|---|---|---|
| MMR | | | | | |
| MR <sup>4</sup> | | | | | |

# **Regained MMR**

Table 12: Results for relapsed patients who regained MMR

| Group | No. of relapsed patients | No. of patients<br>who regained<br>MMR on<br>resumption | % of patients<br>who regained<br>MMR on<br>resumption | 90%<br>Confidence<br>Interval |
|---|---|---|---|---|
| MMR | | | | |
| MR <sup>4</sup> | | | | |

# Molecular relapse-free survival

Table 13: Results for molecular relapse-free survival

| | MMR<br>N = | MR <sup>4</sup><br>N = | Total<br>N = |
|---|---|---|---|
| Molecular relapses, n(%) | | | |
| Median time to molecular relapse in months (IQR) - "if estimable" | | | |

Figure 3: Kaplan-Meier plot for molecular relapse-free survival (Example)



Table 14: Results for molecular relapse-free survival according to MR<sup>4.5</sup> status

| | MMR – MR <sup>4.5</sup><br>N = | MMR – not MR <sup>4.5</sup><br>N = | MR <sup>4</sup> - MR <sup>4.5</sup><br>N= | MR <sup>4</sup> – not MR <sup>4.5</sup><br>N= |
|---|---|---|---|---|
| Molecular relapses, n(%) | | | | |
| Median time to molecular relapse in months (IQR) - "if estimable" | | | | |

Figure 4: Kaplan-Meier plot for molecular relapse-free survival according to MR<sup>4.5</sup> status (Example)



# **Progression-free Survival**

Table 15: Results for progression-free survival

| | MMR<br>N = | MR <sup>4</sup><br>N = | Total<br>N = |
|---|---|---|---|
| Progressions/deaths (first occurrence), n(%) | | | |
| Median time to progression/death in months (IQR) - "if estimable" | | | |

Figure 6: Kaplan-Meier plot for progression-free survival (Example)



## **Overall Survival**

**Table 16: Results for overall survival** 

| | MMR<br>N = | MR <sup>4</sup><br>N = | Total<br>N = |
|---|---|---|---|
| Deaths from any cause, n(%) | | | |
| Median time to death in months (IQR) "if estimable" | | | |

Figure 6: Kaplan-Meier plot for overall survival (Example)



## **Event-free survival**

Table 17: Results for event-free survival

| | MMR<br>N = | MR <sup>4</sup><br>N = | Total<br>N = |
|---|---|---|---|
| Losses of MMR / progressions to AP/BC / deaths (first occurrence), n(%) | | | |
| Median time to death in months (IQR) "if estimable" | | | |

Figure 7: Kaplan-Meier plot for event-free survival (Example)



# Time to MMR recovery

Table 18: Results for time to MMR recovery

| | MMR<br>N = | MR <sup>4</sup><br>N = | Total<br>N = |
|---|---|---|---|
| MMR recoveries, n(%) | | | |
| Median time to MMR recovery in months (IQR) "if estimable" | | | |

Figure 8: Cumulative incidence plot for time to MMR recovery

# MR<sup>4.5</sup> prior study entry

Table 19: Proportion of MMR and MR<sup>4</sup> in confirmed MR<sup>4.5</sup> prior entering the study

| Group | No. of patients<br>MR <sup>4.5</sup> prior study<br>entry | % of patients<br>MR <sup>4.5</sup> prior<br>study entry | 90%<br>Confidence<br>Interval |
|---|---|---|---|
| MMR | | | |
| MR <sup>4</sup> | | | |

# **Quality of Life and TKI related symptoms**

Figure 9: EQ-index score profile over time (example)

EQ-index Score range: 0 – 100 (0: worst possible score, 100: best possible score)



Figure 9: EQ-VAS score profile over time (example)

EQ-VAS Score range: 0 – 100 (0: worst possible score, 100: best possible score)



Figure 11: Mean FACT-BRMTOI score profile over time (example)

FACT-BRMTOI Score range: 0 – 106 (0: worst possible score, 106: best possible score)



Figure 12: Mean FACT-G score profile over time (example)

FACT-G Score range: 0 – 106 (0: worst possible score, 106: best possible score)



Figure 13: FACT-BRM total score profile over time (example)

FACT –BRM Total Score range: 0 – 160 (0: worst possible score, 160: best possible score)



Table 20: Joint longitudinal and survival modelling of QoL data.

| Component | Parameter | Estimate | SE | 90% Confidence<br>interval |
|---------------|-----------|----------|----|----------------------------|
| | Factor 1 | | | |
| Longitudinal | Factor 2 | | | |
| Model | Factor 3 | | | |
| | ••• | | | |
| | Factor 1 | | | |
| Failure Model | Factor 2 | | | |
| railure Model | Factor 3 | | | |
| | ••• | | | |
| Association | ••• | | | |
| Variance | ••• | | _ | |
| Parameters | | | | |

Figure 14: Kaplan Meier plot to show overall survival and integrated QoL utility over time.

Table 21: Number of Patient with TKI related symptoms.

| Time<br>point<br>(month) | Group | Rash | Diarrhoea | Nausea | Scalp<br>irritation | Periobital<br>oedema | Hair<br>thinning | Lethargy | Other | 3+ CTCAE<br>Grade |
|---|---|---|---|---|---|---|---|---|---|---|
| Baseline | MMR | | | | | | | | | |
| Daseille | MR4 | | | | | | | | | |
| 1 | MMR | | | | | | | | | |
| 1 | MR4 | | | | | | | | | |
| 2 | MMR | | | | | | | | | |
| 2 | MR4 | | | | | | | | | |
| 2 | MMR | | | | | | | | | |
| 3 | MR4 | | | | | | | | | |
| | MMR | | | | | | | | | |
| 6 | MR4 | | | | | | | | | |
| 0 | MMR | | | | | | | | | |
| 9 | MR4 | | | | | | | | | |
| | ••• | | | | | | | | | |

Figure 12: Number of Patient with TKI related symptoms over time (radar plot).

# 5.9. Analysis of safety & tolerability

The number and percentage of patients reporting a Serious Adverse Event (SAE) lead to study discontinuation will be summarised by group.

Table 21: N (%) Patients withdrawing due to SAE

| | MMR | MR <sup>4</sup> |
|-------------------|-----|-----------------|
| N (%) | | |
| Mean SAEs/patient | | |

The number of patients reporting a serious adverse event will be summarised by group and CTCAE preferred term.

**Table 22: Aggregated Serious Adverse Event** 

| CTCAE category | CTCAE short name | MMR | MR <sup>4</sup> |
|----------------|------------------|-----|-----------------|
| YYYY | aaaaa | | |
| | bbbbb | | |
| | ccccc | | |
| XXXX | ааааа | | |
| | bbbbb | | |
| | ccccc | | |

Table 23: Line Listing of Grade 3+ Serious Adverse Events

| Patient No | Group | CTCAE<br>Event<br>Name | CTCAE<br>Grade | Onset<br>Date | Offset<br>Date | Outcome |
|---|---|---|---|---|---|---|

# **FINAL REPORT PLAN SIGN-OFF SHEET**

This confirms approval of the Final report plan version 2 for DESTINY

| Trial statistician: | | |
|------------------------|--------------|------|
| Signature | She Gas | |
| Date | 17/07/2019 | |
| Reviewing statisticia | n: | |
| Signature | 2 | |
| Date | 17/07/2019 | |
| Chief Investigator: | | |
| Signature | 17/07/2019. | |
| Date | 17/07/2019. | |
| Chair of Trial Steerin | g Committee: | |
| | - TE | |
| Signature | | <br> |
| Date | 17/07/2019 | 1 16 |

Add: Retain Original Copy of Final Report Plan & Sign-off sheet in appropriate sections of Statistics File

Keep a scanned copy of each in corresponding electronic folder





# **FINAL STATISTICAL REPORT SIGN-OFF SHEET**

| Programming and Reporting Checklist for DESTINY Final statistical report | TS | RS |
|---|---|---|
| Programming | | |
| Has the relevant analysis plan been written and signed off | | |
| Timescales agreed for database lock, data download into R/Stata/SAS etc, analysis and dissemination | | |
| Have MACRO Queries been created to supply data needed for each table /figure in Report | | |
| Have you checked that the data have been read into SAS/Stata correctly | | |
| Have all SAS/Stata/etc analysis programs been listed in the relevant index? | | |
| Have all SAS/Stata/etc analysis programs been risk-assessed, with appropriate review & sign-off in the validation log | | |
| Have the numbers in the tables been checked against the relevant SAS/Stata output | | |
| Report | | |
| Pagination correct | | |
| Open meeting section clearly distinct from closed section (DMC Report) | | |
| All tables/graphs stipulated in Report Plan/subsequent amendments are present/accounted for | | |
| Layout & formatting acceptable (percentages as a whole number, means to 1 d.p. more than unit of measurement) | | |
| Table rows/columns labelled clearly, with units | | |
| Graph axes labelled clearly, with units | | |
| All accompanying text consistent with presented results | | |
| Has report been reviewed and signed off by statistical lead? | | |

This confirms approval of the Final Statistical Report for DESTINY

Signed (TS)
Date
Signed (RS)
Date

Retain Original Copy of Report & Sign-off sheet in appropriate sections of Statistics File

Keep a scanned copy of each in corresponding electronic folder